CLINICAL TRIAL: NCT05485168
Title: Combined Effects of Sequential Variety and Portion Size on Meal Intake of Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FoodVariety104
Record Dates: First submitted 2022-07-28; First posted 2022-08-03 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequential Variety, Small Portion (Experimental): 3 different foods served in a small portion in 3 successive courses
  Interventions: Other: Sequential Variety; Other: Small Portion
- Sequential Variety, Large Portion (Experimental): 3 different foods served in a large portion in 3 successive courses
  Interventions: Other: Sequential Variety; Other: Large Portion
- Single-Food, Small Portion (Experimental): 1 food served in a small portion in 3 successive courses
  Interventions: Other: Single-Food; Other: Small Portion
- Single-Food, Large Portion (Experimental): 1 food served in a large portion in 3 successive courses
  Interventions: Other: Single-Food; Other: Large Portion

INTERVENTIONS:
Other: Sequential Variety — 3 different foods served in 3 successive courses
  Arms: Sequential Variety, Large Portion; Sequential Variety, Small Portion
Other: Single-Food — 1 food served in 3 successive courses
  Arms: Single-Food, Large Portion; Single-Food, Small Portion
Other: Small Portion — Small meal portion size
  Arms: Sequential Variety, Small Portion; Single-Food, Small Portion
Other: Large Portion — Large meal portion size
  Arms: Sequential Variety, Large Portion; Single-Food, Large Portion

SUMMARY:
The primary purpose of this study is to investigate the combined effects of sequential meal variety and portion size on food intake at a meal. Additionally, other individual characteristics will be examined for their influence on the effects of simultaneous variety and portion size on meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to travel to Penn State University Park campus weekly for meals
* Be fully vaccinated against COVID-19
* Be a woman 20 - 65 years old
* Regularly eat 3 meals/day
* Be willing to refrain from drinking alcohol the day before and during test days
* Have a body mass index between 18.0 and 35.0 kg/m*m
* Be willing to refrain from eating after 10 pm the evening before test sessions
* Be willing to participate in all study procedures

Exclusion Criteria:

* Must not be a smoker
* Must not be an athlete in training
* Must not be pregnant or breastfeeding at the time of screening
* Must not have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Must not dislike or be unable to eat the test foods (because of allergies, intolerance, or dietary restrictions)
* Must not have a high variability in liking of the test foods
* Must not be currently dieting to gain or lose weight
* Must not have a health condition that affects appetite
* Must not have participated in a similar study in our lab in the past year
* Must not be a student, faculty, or staff member in nutritional sciences or psychology

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Change in intake by weight | Weeks 1, 2, 3, 4
  Weight (grams) of all meal components consumed
Change in energy intake | Weeks 1, 2, 3, 4
  Energy intake (kilocalories) of all meal components consumed, calculated from weight and energy density

SECONDARY OUTCOMES:
Change in bite count | Weeks 1, 2, 3, 4
  The number of bites of food during the meal
Change in active eating time | Weeks 1, 2, 3, 4
  Duration of the time spent eating in minutes
Change in mean eating rate | Weeks 1, 2, 3, 4
  Mean food intake per minute (grams/minute), calculated by dividing meal food intake by meal duration
Change in mean bite size | Weeks 1, 2, 3, 4
  Mean food intake per bite (grams/bite), calculated by dividing meal food intake by bite count
Change in sip count | Weeks 1, 2, 3, 4
  The number of sips of water during the meal
Change in mean drinking rate | Weeks 1, 2, 3, 4
  Mean water intake per minute (grams/minute), calculated by dividing meal water intake by meal duration
Change in mean sip size | Weeks 1, 2, 3, 4
  Mean water intake per sip (grams/sip), calculated by dividing meal water intake by sip count
Change in switching between bites and sips | Weeks 1, 2, 3, 4
  The number of switches between bites and sips during the meal
Change in rating of pleasantness of the taste of food samples | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all pleasant (0 mm) to extremely pleasant (100 mm). This will be used to calculate Sensory-Specific Satiety
Change in rating of desire to eat food samples | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all strong (0 mm) to extremely strong (100 mm), in answer to "How strong is your desire to eat [this food] right now?". This will be used to calculate Sensory-Specific Satiety.
Change in rating of hunger | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all hungry (0 mm) to extremely hungry (100 mm)
Change in rating of thirst | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all thirsty (0 mm) to extremely thirsty (100 mm)
Change in rating of nausea | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all nauseated (0 mm) to extremely nauseated (100 mm)
Change in rating of fullness | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from not at all full (0 mm) to extremely full (100 mm)
Change in rating of prospective consumption | Weeks 1, 2, 3, 4
  Measured on a 100-mm visual analogue scale ranging from nothing at all (0 mm) to a large amount (100 mm), in answer to "How much food do you think you could eat right now?".

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No